CLINICAL TRIAL: NCT02398344
Title: THE IMMEDIATE EFFECT OF ELECTRICAL STIMULATION TRANSCRANIAL DIRECT CURRENT (tDCS) ON CARDIORESPIRATORY PARAMETERS IN HEMIPARETICS ADULTS PATIENTS DUE TO STROKE
Brief Title: tDCS Immediate Effect on Cardiorespiratory Parameters in Hemiparetics Adults Patients Due to Stroke.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Catarina Novaes Sousa Bertani, Catarina Novaes Sousa Bertani, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: '738.356
Record Dates: First submitted 2015-02-21; First posted 2015-03-25 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1- tDCS ACTIVE (Experimental): 1. Transcranial stimulation ( tDCS ) will be administered using Tct Research 1 CH tdcs Simulator model 101. tDCS will be performed for 20 minutes, intensity 2mA With Simulator anodic electro stimulation from bloodstream on right and left temporal cortex region (T3 area) and cathodic position in contralateral supraorbital region to anode (Fp2), associated Cardiac Frequency Variability (HRV) as measured by spectral analysis by spectral analysis Polar RS800 cx.
  Interventions: Device: tDCS active
- 2- tDCS SHAM (Experimental): Placebo tDCS will be administered using Tct Research 1 CH tdcs Simulator model 101 and will follow the same procedures as active tDCS active, but the tDCS device will only be switched on for 30 seconds.
  Interventions: Device: tDCS Sham

INTERVENTIONS:
Device: tDCS active — Transcranial direct current stimulation (tDCS) the active tDCS and placebo will be applied to the temporal cortex (T3) associated Cardiac Frequency Variability (HRV).
  Arms: 1- tDCS ACTIVE
Device: tDCS Sham — Active stimulation application time or placebo 20 minutes. In all sham stimulation, electrode placement procedures will also be performed like the procedures with anodic tDCS, the left and right temporal cortex, however, the stimulator is turned on for 30 seconds only, and the patient will be told that he will feel a slight initial tingling, but it will reduce, disappear or remain during the 20 minutes of application. Thus, individuals will feel it initially, but receive no stimulation in the remaining time. This procedure is a valid form of control in challenge studies transcranial direct current ³³. The equipment itself has a sham configuration.
  Arms: 2- tDCS SHAM

SUMMARY:
Previous studies found important function of brain in exercises regulation on healthy and athlete patients and this studies showed not invasive stimulation on temporal cortex brain, induces electrics field to insula cortex, in addition modulate autonomic nervous system cognition efforts during submaximal (maximal hight frequency) and maximal exercises. Measure immediate effects of transcranial stimulation in bloodstream (tDCS) anodic on right and left temporal cortex in the cardiorespiratory parameters (functional capacity, perception of efforts and modulation of autonomic nervous system) in patients with hemiparesis due stroke. Methods and Material: It Is a clinical trial, controlled and Double blind, using 30 adult patients with stroke sequel, like roam. Evaluation will be hemodynamic measure data such as: Heart Rate, Respiratory Rate, Blood Pressure, Lung Capacity Vital and assessment of the Autonomic Nervous System, before and after anodic electro stimulation from bloodstream on right and left temporal cortex region (T3 area) and cathodic position in contralateral supraorbital region to anode (Fp2). On temporal cortex will be applied of 2mA during stimulation of 20 minutes. Sham stimulation all electrodes Will be used. The stimulator turns on for 30 seconds. Results: The primary results will analyze cardiac frequency before and after tDCS and second step will assess the travelled distance on walking test for 6 minutes with and without tDCS and compare these respiratory reviews results with stroke gravity.

DETAILED DESCRIPTION:
This is a clinical protocol, randomized, crossover, double-blind (patient and data analyst) will be held. The study protocol is registered in clinicalTrials.gov - NCT02398344.

Methods

Individuals with AVE will be recruited from the physical therapy clinics of the Universidade Nove de Julho - Sao Paulo, Brazil. The participants will be recruited and selected based on the following eligibility criteria:

Sample size Sample of 20 the participants (05 participants in each level of motor impairment - mild, moderate, marked and severe) will taken. This value will assumed, based on studies of Okano et al.²⁰ evaluating HRV after tDCS in 10 athletes and Vandermeeren et al.²⁶ that evaluated the effect of tDCS over the cardiorespiratory system in 30 healthy individuals.

As the primary outcome will considered the heart rate variability, validated for the population of adults with hemiparesis after a stroke and a variable considered secondary outcome, by correlating the functional capacity with the severity of the stroke, the 6-minute walk test, considering the cardiorespiratory fitness and the patient's mobility before and after the application of tDCS and correlate whether there are differences on the immediate effect of tDCS applied in both cerebral hemispheres (right and left).

Procedures Initially, participants will be screened at University Nine July physical therapy clinics at São Paulo. Individuals who meet the eligibility criteria will be invited to participate in the study, being included after agreement by signing the Instrument of Consent.

The following description of the evaluation procedures:

Identification form: After screening, an identification sheet of the selected volunteers will be filled in, containing the following information: name, date of birth, age (years and months), topographic diagnosis of stroke, classification of the type of stroke (hemorrhagic or ischemic), weight (kg), height (cm), blood pressure (BP), classification of functional severity according to Fulg Meyer ²⁷ (Mild, Moderate, marked and severe) time since injury, area of committed member, carried out therapies and how long, muscle strength of the paretic body side according to Kendall et al. ²⁸ and Ashworth ²⁹.

Functional Mobility Scale: This scale will be used for screening, in order to assess how the individual moves in the environment to achieve their interaction in everyday life with family and the social environment. The FMS provides scores in three different lengths (5m, 50m and 500m), relating to mobility at home, school and community. The classification is performed according to the patients needs in assistance to movement and according to the distance ²⁵. The included patient should wander at least 50 m.

All data will be recorded on a card and then the patients will informed about the experimental procedures, including previous recommendations to each test: have a light meal in the days of the tests; abstain from caffeine and alcohol intake and / or smoking, avoid moderate or excessive effort the day before and on test day, have a good night's sleep and present ourself in comfortable clothes and shoes that allow good mobility.

Pulmonary function tests: spirometry evaluation EasyOne Plus Diagnostic Sprometry System® in order to identify the presence of lung function changes measured by forced expiratory volume in the first second (FEV1), forced vital capacity (FVC), peak flow expiratory (PEF) and FEV1 / FVC ratio, according to the criteria of the American Thoracic Society ³⁰. Spirometric indices will be presented in absolute terms and as a percentage of the reference values. Volunteers must complete at least three acceptable and reproducible forced expiratory maneuvers.

Respiratory muscle strength: Respiratory muscle strength will be obtained through maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP), which measures the inspiratory and expiratory muscle strength, respectively, and will be obtained by the method of Black & Hyatt³¹. In order to accomplish these steps, it uses a scaled manometer in cm H2O, with an operating range of ± 300 cmH2O adapter equipped with nozzles and containing a safety valve through a bore, 2mm in diameter, in order to prevent increased pressure in the oral cavity generated exclusively by facial²⁴ muscle contraction. The MIP is obtained by a maximal inhalation maneuver starting from a maximum expiration and MEP obtained by a maximum exhalation maneuver starting from maximum inspiration. Each maneuver will be maintained for a minimum of two to three seconds. The MIP and MEP performed three times for each patient, and, for analysis, will count the highest value obtained ³².

FulgMeyer scale (EFM) - The motor impairment assessment instruments measure the level of motor recovery of hemiplegic patients, highlighting the motor test procedure in Hemiplegia. The proposed measures in the FSM are based on neurological examination and sensory-motor activity of upper and lower limbs in order to identify selective and synergistic activity patterns of patients who suffered strokes. This scale was constructed following the hypothesis that restoration of motor function in hemiplegic patients follow a defined course. It is represented by a three-point ordinal scale that is applied in every item: 0- can not be performed, partially performed 1- and 2 - fully realized. The total of this scale is 100 points for normal motor function, where the maximum score for the upper end is 66 and the lower 34. The motor evaluation includes measurement of motion, coordination and reflex activity of shoulder, elbow, wrist, hand, hip, knee and ankle determining a score according to the motor impairment level, where less than 50 points indicates a severe motor impairment; 85-95 moderate; 50-84 remarkable and 96-99 light ²⁷.

Analysis of heart rate variability (HRV):

The Heart rate variability will be analyzed in four stages:

1. Resting 01: The heart rate (HR) is captured by means of a heart rate monitor (RS800 CX) with online data transmitted to a computer, over a period of 10 minutes of rest. Individuals will be instructed to remain recumbent for 10 minutes, avoiding any activity and without sleep, after this examination the patient will remain in the sitting position posture for over 10 minutes following the same guidelines given above.
2. In exercise: After the initial 20 minutes of rest, the patient will start the six-minute walk test. The FC will be collected through the same heart rate monitor throughout the walk test, as well as in post exercise recovery (for 2minutes). In this recovery the patient will remain in the sitting position, and will be instructed to not verbalize and not move during the evaluation.
3. Electrical stimulation by direct current (Home): After the walk (6MWT) and the recovery of hemodynamic parameters to baseline parameters, stimulation with tDCS in sitting position posture starts, and during stimulation HR will be collected.
4. 6 minute walk test 02: After finishing the tDCS, the patient should again perform the 6MWT through the same guidelines of the American Thoracic Society ³⁰, assessing the FC.

After the test there will be given a continuity of HRV analysis for 2 minutes with the patient in the sitting position, without verbalizing and without moving , in order to analyze the behavior of the autonomic nervous system.

6-minute walk test - a reliable measure for assessing physical fitness and functional mobility ³⁰. The test quantifies in meters the distance traveled by the individual in six minutes. It is performed in accordance with the guidelines established by the American Thoracic Society ³⁰.

During the walk test the patient will be told to stop if he feels bad, there will always be a researcher on the side to avoid possible falls during the test run and will be monitored by the oximeter (More Fitness MF-417®).

2.5.1. Stimulation procedures transcranial direct current The transcranial electrical stimulation DC (tDCS) will be performed with a tag device 1 CH Tct Research tDCS Simulator model 101® by means of two surface sponge electrodes , (non-metallic) 5-7 cm2 in humidified saline, with a 2mA current.

Individuals will be submitted to four experimental conditions, and the order distributed by randomization through manila envelopes.

1. tDCS anode on the left temporal cortex (T3) and cathode on the contralateral supraorbital region;
2. tDCS sham on left temporal cortex (T3) and cathode on the above-orbitalcontralateral region;
3. tDCS anode on the right temporal cortex (T4) and cathode on the contralateral supraorbital region;
4. tDCS sham on right temporal cortex (T4) and cathode on the contralateral supra orbital region.

Protocol 1 and 2: The anode electrode will be positioned on the left temporal cortex (T3), located 40% of the distance from the left side of Cz point following the international 10-20 system electroencephalogram and the cathode electrode on the region supra orbital contralateral to the anode.

Protocol 3 and 4: The anode electrode will be positioned on the right temporal cortex (T4) and cathode positioned on the left supraorbital region.

Active stimulation application time or placebo 20 minutes. In all sham stimulation, electrode placement procedures will also be performed like the procedures with anodic tDCS, the left and right temporal cortex, however, the stimulator is turned on for 30 seconds only, and the patient will be told that he will feel a slight initial tingling, but it will reduce, disappear or remain during the 20 minutes of application. Thus, individuals will feel it initially, but receive no stimulation in the remaining time. This procedure is a valid form of control in challenge studies transcranial direct current ³³. The equipment itself has a sham configuration.

According to Okano et al. ²⁰, before receiving any of the experimental conditions (transcranial direct-current stimulation (anodic or sham), individuals must rest for a period of 10 minutes (sitting comfortably), so that the cardio respiratory variables return to baseline measurements.

The two study conditions (anodic stimulation and sham) will be performed with an interval of 48 hours ³⁴ and always in the same period of the day.

Protective measures to subjects Patients will be exposed to minimal risk during the search, trying to be controlled at all times by the researcher, who will accompany and monitor all cardiorespiratory changes, giving support if the patient has imbalance or discomfort, and interrupting the action immediately if necessary.

ELIGIBILITY:
Inclusion Criteria:

* 30 individuals wich hemiparesis stemming from a stroke;
* Rating of Functional Mobility Scale levels (FMS- functional mobility scale)
* Walking at least 50 meters (GRAHAN et al. 2004); Science signature in consent term exempt and enlightened (TCLE) .

Exclusion Criteria:

* Positive Cutoff to cognitive wastage screening (mental mini) - Visual commitment may intervene in tests achievement;
* Cardiac vast problems and use of pacemaker;
* Contraindication of tDCS application (history of recurrent seizures, recurrent epilepsy and brain tumor in stimulation site);

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cardiac Frequency Variability (HRV) as measured by spectral analysis by Polar RS800 cx. | 1 years
  Individuals with right lesion, after anodal tDCS wolf T3 (healthy): BF (p=0,32), AF(p=0,88), LF/HF (p=0,18); tDCS in T4 (injured): BF (p=0,90), AF (p=0,19) and LF/HF (p=0,29). Individuals with left foot injury, tDCS in wolf T3 (injured) BF (p=0,15), AF (p=0,12) and LF/HF (p=0,81) and tDCS wolf T4 (healthy): BF (p=0,89), AF (p=0,18) and LF/HF (p=0,34).

CONTACTS AND LOCATIONS:
Overall Officials: Catarina NS Bertani, specialist, Principal Investigator — University Nive July
Locations (1):
- University of Nove de Julho, São Paulo, São Paulo, Brazil